CLINICAL TRIAL: NCT03335371
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Multiple-Dose, Adaptive Study Assessing the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of TTP399 in With Adult Patients Type 1 Diabetes Mellitus
Brief Title: Evaluation of TTP399 in Patients With Type 1 Diabetes
Acronym: SimpliciT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TTP399-203; JDRF#2-IND-2018-500 (Other: JDRF International)
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — TTP399

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TTP399 400 mg (Experimental)
  Interventions: Drug: TTP399
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: TTP399 — Phase 1: Participants will receive TTP399 administered orally up to 1200 mg taken once daily for 7 days
  Arms: TTP399 400 mg
Drug: TTP399 — Phase 2: Participants will receive TTP399 administered orally 800 mg taken once daily for 12 weeks
  Arms: TTP399 400 mg
Drug: Placebo Oral Tablet — Phase 2: Participants will receive Placebo oral tablets for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TTP399 in Type 1 diabetics. This study will be in 2 phases: phase 1 will evaluate the safety of different TTP399 dosage regimens over 1 week of daily dosing. Phase 2 will evaluate the safety and efficacy of a TTP399 dosing regimen over 12 weeks of daily dosing.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with T1DM, confirmed diagnosis prior to 40 years of age and a diagnosed for minimum of 1 year.
* Type 1 diabetics using either continuous subcutaneous insulin infusion (with lispro or aspart) or multiple daily doses of insulin
* Willing to use adequate contraception
* No major surgeries or significant injuries within the past year and without an active infection.

Exclusion Criteria:

* Diagnosis of T2DM, severely uncontrolled T1DM, maturity-onset diabetes of the young, insulin-requiring T2DM, other unusual or rare forms of diabetes mellitus, diabetes resulting from a secondary disease
* Receipt of an investigational product within 30 days of the Screening Visit or any therapeutic protein or antibody within 90 days prior to Screening Visit or any previous treatment with TTP399.
* Living in the same household or related to another participant in this study.
* Two severe episodes of hypoglycemia that required assistance by a third party within 3 months of Screening Visit
* Use of antidiabetic medications other than insulin 3 months prior to Screening Visit, systemic corticosteroids 1 month prior to Screening Visit, weight loss medication 2 weeks prior to Screening Visit, and antipsychotic medications 3 months prior to Screening Visit.
* Participation in any formal weight loss program or contemplating such therapy during the trial.
* Recent history of use of non-prescribed controlled substances or illicit drugs.
* Current alcoholism or a history of excessive alcohol consumption within 2 years prior to screening
* History or presence of symptomatic autonomic neuropathy or chronic gastrointestinal disease.
* Personal history of long QT syndrome.
* Blood donation of approximately 1 pint (500 mL) within 8 weeks before Screening Visit
* History of hemolytic anemia or chronic transfusion requirement.
* History of cancer, other than non-melanoma skin cancer or uterine cervical cancer that required therapy in the past 5 years.
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Valcarce, Ph.D., Study Director — vTv Therapeutics, LLC
Locations (15):
- United States (15):
  - USC Westside Center for Diabetes, Beverly Hills, California
  - AMCR Institute, Escondido, California
  - University of Colorado Barbara Davis Center, Aurora, Colorado
  - Atlanta Diabetes Associate, Atlanta, Georgia
  - Rocky Mountain Diabetes Center, Idaho Falls, Idaho
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - UNC Diabetes Care Center, Chapel Hill, North Carolina
  - Duke University Diabetes Research Clinic, Durham, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Intend Research, Norman, Oklahoma
  - Dallas Diabetes Research Center, Dallas, Texas
  - University of Washington Medicine Diabetes Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein KR, Freeman JLR, Dunn I, Dvergsten C, Kirkman MS, Buse JB, Valcarce C; SimpliciT1 research group. The SimpliciT1 Study: A Randomized, Double-Blind, Placebo-Controlled Phase 1b/2 Adaptive Study of TTP399, a Hepatoselective Glucokinase Activator, for Adjunctive Treatment of Type 1 Diabetes. Diabetes Care. 2021 Apr;44(4):960-968. doi: 10.2337/dc20-2684. Epub 2021 Feb 23. PMID 33622669

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 110 participants were randomized to the study groups: Sentinel, Part 1, and Part 2. Sentinel participants were the same participants throughout the dose levels.
Groups:
- Sentinels: Sentinel: Participants who received TTP399 400 mg administered orally once daily for 1 week per dose level.
  Period 1: 400 mg TTP399 administered Period 2: 800 mg TTP399 administered Period 3: 1200 mg TTP399 administered
- Part 1 TTP399 800 mg: TTP399 Part 1: Participants who received TTP399 800 mg administered orally once daily for 12 weeks with a 1-week follow-up after the last dose was administered.
- Part 1 Placebo: Placebo Part 1: Participants who received placebo tablets administered orally once daily for 12 weeks with a 1-week follow-up after the last dose was administered.
- Part 2 TTP399 800 mg: TTP399 Part 2: Participants who received TTP399 800 mg administered orally once daily for 12 weeks with a 1-week follow-up after the last dose was administered.
- Part 2 Placebo: Placebo Part 2: Participants who received placebo tablets administered orally once daily for 12 weeks with a 1-week follow-up after the last dose was administered.
Period: Overall Study
Arm/Group | Sentinels | Part 1 TTP399 800 mg | Part 1 Placebo | Part 2 TTP399 800 mg | Part 2 Placebo
Started | 5 | 9 | 11 | 40 | 45
Completed | 5 | 9 | 10 | 40 | 43
Not Completed | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Randomization Error | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sentinel participants were the same participants throughout the dose levels. Part 1 is the full analysis set. Part 2 is all randomized subjects who received at least 1 dose of the investigational product.
Groups:
- Sentinel: Sentinel: Participants who received TTP399 400 mg, 800 mg, and 1200 mg administered orally once daily for 1 week per dose level.
- Total: Total of all reporting groups
Arm/Group | Sentinel | Part 1 TTP399 800 mg | Part 1 Placebo | Part 2 TTP399 800 mg | Part 2 Placebo | Total
Number analyzed (Participants) | 5 | 8 | 11 | 40 | 45 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7.4) | 38 (15.71) | 47 (10.10) | 43 (15.26) | 42 (13.26) | 42.5 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8 | 15 | 25 | 56
  Male | 2 | 3 | 3 | 25 | 20 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 8 | 11 | 39 | 43 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 2
  White | 5 | 7 | 11 | 38 | 43 | 104
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 24 (3) | 28 (3.30) | 29 (4.13) | 28 (4.16) | 28 (3.76) | 28 (3.8)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent HbA1c in blood] | 6.9 (0.7) | 7.20 (0.42) | 7.36 (0.41) | 7.66 (0.56) | 7.52 (0.59) | 7.45 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: To evaluate the change in glycosylated hemoglobin (HbA1C) in Part 1 and Part 2 participants following multiple-day dosing (at 12 weeks) in subjects with T1MD. Sentinel participants were not evaluated for a change in HbA1C.
Time Frame: Baseline (Day 1) to Week 13
Population: Part 1 and Part 2 populations are the full analysis of randomized subjects. Sentinel participants were not evaluated for a change in HbA1C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Part 1 Placebo: Placebo Part 1: Participants will receive Placebo oral tablets for 12 weeks
- Part 1 TTP399 800 mg: TTP399 Part 1: Participants will receive TTP399 administered orally 800 mg taken once daily for 12 weeks
- Part 2 Placebo: Placebo Part 2: Participants will receive Placebo oral tablets for 12 weeks
- Part 2 TTP399 800 mg: TTP399 Part 2: Participants will receive TTP399 administered orally 800 mg taken once daily for 12 weeks
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 45 | 40
percent change | 0.08 (0.2) | -0.60 (0.2) | 0.07 (0.06) | -0.14 (0.06)
Statistical Analysis 1: Comparison: Part 2 Placebo vs Part 2 TTP399 800 mg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.39 to -0.04], Standard Deviation 0.087

2. Primary Outcome: Sentinel - Area Under the Concentration Time Curve (AUC)
Description: AUC for Day 1 per dose level (400 mg, 800 mg, and 1200 mg) is AUC from 0 to 9 hours.
Time Frame: Predose, 60, 90, 120, 150, 180, 240, 360 (6hr) and 540min (9hr) after dosing.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Sentinel 400 mg: Sentinel: Participants who received TTP399 400 mg administered orally once daily for 1 week per dose level.
- Sentinel 800 mg: Sentinel: Participants who received TTP399 800 mg administered orally once daily for 1 week per dose level.
- Sentinel 1200 mg: Sentinel: Participants who received TTP399 1200 mg administered orally once daily for 1 week per dose level.
Arm/Group | Sentinel 400 mg | Sentinel 800 mg | Sentinel 1200 mg
Number analyzed (Participants) | 5 | 5 | 5
ng*h/mL | 1778 (992) | 1482 (341) | 4848 (2663)

3. Primary Outcome: Sentinel - Maximum Drug Concentration (Cmax)
Time Frame: Predose, 60, 90, 120, 150, 180, 240, 360 (6hr) and 540min (9hr) after dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sentinel 400 mg | Sentinel 800 mg | Sentinel 1200 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 645 (219) | 813 (129) | 2038 (1415)

4. Secondary Outcome: Percent Change From Baseline Time in Target Glycemic Range (70-180 mg/dL)
Description: To evaluate the change from baseline time in target range (24 hour)
Time Frame: Baseline (Day 1) to Week 12
Population: Part 1 is the full analysis set. Part 2 is all randomized subjects who received at least 1 dose of the investigational product.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
percent change | -8 (10) | -3 (8) | -7 (14.0) | 0.50 (16)

5. Secondary Outcome: Percent Change From Baseline Time in Hypoglycemia (< 54 mg/dL)
Description: To evaluate the change from baseline time in hypoglycemia (< 54 mg/dL)
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
percent change | -0.1 [-2 to 2] | -0.1 [-3 to 0] | -0.5 [-8 to 8] | -0.5 [-8 to 22]

6. Secondary Outcome: Percent Change From Baseline Time in Hypoglycemia (< 70 mg/dL)
Description: To evaluate the change from baseline time in hypoglycemia (< 70 mg/dL)
Time Frame: Baseline (Day 1) to Week 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
percent change | -1 (3) | -1 (3) | -2 (5) | -2 (8)

7. Secondary Outcome: Percent Change From Baseline Time in Hyperglycemia (>180 mg/dL)
Description: To evaluate the change from baseline time in hypoglycemia (>180 mg/dL)
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Part 1 Placebo: Placebo Part 1: Participants will receive Placebo oral tablets for 12 week
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
percent change | 9 (12) | 5 (8) | 10 (17) | 1 (18)

8. Secondary Outcome: Percent Change From Baseline Time in Hyperglycemia (>250 mg/dL)
Description: To evaluate the change from baseline time in hypoglycemia (>250 mg/dL)
Time Frame: Baseline (Day 1) to Week 12
Population: Time in hypoglycemia >250mg/dL was only evaluated in Part 2 of the study. Part 2 is all randomized subjects who received at least 1 dose of the investigational product.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 43 | 38
percent change | 6 (11) | 2 (12)

9. Secondary Outcome: Percent Change From Baseline in Total Daily Insulin Use
Description: To evaluate the percent change from baseline in total daily insulin use at week 12.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
percent change | -0.1 (8.7) | -1.7 (14.7) | -1.6 (16) | -7.6 (10.1)

10. Secondary Outcome: Change From Baseline in Bolus Insulin Use
Description: To evaluate the change from baseline in bolus insulin use
Time Frame: Baseline (Day 1) to Week 12
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
units/kg/day | -5.9 (17.5) | -1 (31.8) | -3.9 (28.4) | -8.4 (22.7)

11. Secondary Outcome: Change From Baseline in Basal Insulin Use
Description: To evaluate the change from baseline in basal insulin use
Time Frame: Baseline (Day 1) to Week 12
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Part 1 Placebo | Part 1 TTP399 800 mg | Part 2 Placebo | Part 2 TTP399 800 mg
Number analyzed (Participants) | 11 | 8 | 43 | 38
units/kg/day | 4.4 (7.7) | -2.3 (10.3) | -0.5 (11.6) | -5.4 (7.1)

12. Primary Outcome: Sentinel - Time to Maximum Concentration (Tmax)
Time Frame: Predose, 60, 90, 120, 150, 180, 240, 360 (6hr) and 540min (9hr) after dosing.
Measure: Median (Full Range); unit: hour
Arm/Group | Sentinel 400 mg | Sentinel 800 mg | Sentinel 1200 mg
Number analyzed (Participants) | 5 | 5 | 5
hour | 1.5 [1.5 to 2.5] | 1.5 [1.5 to 2.0] | 2.5 [1.5 to 3.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were those reported at baseline up to 12 weeks (±3) days after the last dose. Unresolved AEs were followed up by the investigator for as long as medically indicated. Sentinel group reported at baseline up to 28 days after the last dose.
Description: The safety analysis set includes all patients who received at least one dose of study medication. Sentinel participants were the same participants throughout the dose levels.
Groups:
- Placebo (Part 1 and Part 2): Placebo Part 1 and Part 2: Participants will receive Placebo oral tablets for 12 weeks
- TTP399 800 mg (Part 1 and Part 2): TTP399 Part 1 and TTP399 Part 2: Participants will receive TTP399 administered orally 800 mg taken once daily for 12 weeks
Arm/Group | Sentinel 400 mg | Sentinel 800 mg | Sentinel 1200 mg | Placebo (Part 1 and Part 2) | TTP399 800 mg (Part 1 and Part 2)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/56 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 1/56 | 1/49
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5 | 2/5 | 32/56 | 25/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel 400 mg (N=5) | Sentinel 800 mg (N=5) | Sentinel 1200 mg (N=5) | Placebo (Part 1 and Part 2) (N=56) | TTP399 800 mg (Part 1 and Part 2) (N=49)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel 400 mg (N=5) | Sentinel 800 mg (N=5) | Sentinel 1200 mg (N=5) | Placebo (Part 1 and Part 2) (N=56) | TTP399 800 mg (Part 1 and Part 2) (N=49)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 9 (27) | 5 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Eye Discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03335371/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03335371/SAP_001.pdf